CLINICAL TRIAL: NCT03159520
Title: A Randomised Clinical Trial of Advice Regarding Acupressure or NSAIDs for the Control of Orthodontic Pain
Brief Title: Control of Pain From Braces With Patient Advice Sheets
Acronym: COPPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, David Bearn, Principal Investigator, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017OR02
Record Dates: First submitted 2017-05-14; First posted 2017-05-18 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Orthodontic Appliance Complication
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomised parallel clinical trial
Who Masked: Outcomes Assessor
Masking Description: Not possible to mask due to nature of intervention except for outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advice on acupressure (Active Comparator): Advice sheet on use of acupressure for post orthodontic pain
  Interventions: Behavioral: Advice sheet
- Advice on analgesics (Active Comparator): Advice sheet on use of NSAID analgesics for post orthodontic pain
  Interventions: Behavioral: Advice sheet

INTERVENTIONS:
Behavioral: Advice sheet — Advice on management of post orthodontic pain

SUMMARY:
To compare the analgesic property of acupressure with NSAIDs (Ibuprofen) in controlling pain following orthodontic treatment. This will be achieved by assessing the effectiveness of acupressure in controlling pain and discomfort by measuring the degree of pain relief after bonding of brackets to teeth and placement of initial archwire.

DETAILED DESCRIPTION:
Single centred randomised controlled trial with subjects recruited from a hospital orthodontic outpatient department in Dundee Dental Hospital.

If informed consent is obtained, then the subject details will be delivered to the trial coordinator for randomisation to one of the groups, NSAIDs or acupressure group.

All subjects who are eligible for inclusion will be advised of the nature and purpose of the trial. The total number of subjects recruited will be approximately 36 with the acupressure and NSAID group containing approximately 18 subjects each.

All subjects who meet the inclusion criteria will be informed of the study and written consent sought for their participation. Subjects will be recruited from the new patient clinics and routine treatment waiting list. .

The subjects will be asked to measure the level and duration of pain and discomfort using a pain diary to record their experiences using visual analogue scales (VAS). The pain diary will be completed from 4 hours to 7 days after treatment after the insertion of the first orthodontic aligning archwire.

Intervention Groups In the acupressure group the subjects will be given an advice sheet and advised to use a definitive acupressure point on the back of the hand region to control orthodontic pain.

In the NSAID group the subjects will be given an advice sheet and advised to take Ibuprofen for the orthodontic pain

Pain scores via VAS will be analysed at 4hours, 24 hours, and 7 days after the orthodontic treatment. The VAS consists of a horizontal line, 100 mm in length with descriptive words at each end of the line which act as anchors e.g. no pain, great pain. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks

ELIGIBILITY:
Inclusion Criteria:

* aged 12-25
* malocclusion requiring treatment
* scheduled to begin orthodontic treatment
* requires fixed orthodontic braces on upper and lower teeth.

Exclusion Criteria:

* previous orthodontic treatment
* current use of analgesics
* contraindications to the use of NSAIDs
* previous acupressure experience
* pregnant

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Pain experience | 7 days
  Visual analogue scale

SECONDARY OUTCOMES:
Impact of pain on sleep | 7 days
  Impact of pain on sleep as recorded in pain diary
Impact of pain on eating | 7 days
  Impact of pain on eating as recorded in pain diary
Rescue medication | 7 days
  Need to use rescue medication to manage pain as recorded in pain diary

CONTACTS AND LOCATIONS:
Overall Officials: David R Bearn, BDS, Principal Investigator — University of Dundee
Locations (1):
- Dundee Dental Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No